CLINICAL TRIAL: NCT04357639
Title: Prospective Description Study of the Impact of Long-term Protease Inhibitors in Patients Living With HIV on the Incidence of COVID-19
Brief Title: Impact of Long-term Protease Inhibitors in Patients Living With HIV on the Incidence of COVID-19 ( COVIP )
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Centre Hospitalier Intercommunal Villeneuve St Georges (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVIP
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: HIV Patients
Keywords: Protease inhibitor, antiretroviral drug, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protease inhibitor exposed: HIV patients treated with antiretroviral drugs including a protease inhibitor
  Interventions: Other: No intervention
- Protease inhibitor non exposed: HIV patients treated with antiretroviral drugs without a protease inhibitor
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention: Usual care for nasopharyngeal sampling and blood sampling for COVID-19 detection

SUMMARY:
This is a prospective multicenter cohort study. The question arises as to whether treatment with protease inhibitors (PIs) could have a preventive role for COVID-19 infection, especially since patients living with HIV (PLWHIV) have not been described as more at risk of developing COVID-19 infection.

The aim of our study will therefore be to assess the impact of long-term protease inhibitors in PLWHIV on the incidence of COVID-19.

DETAILED DESCRIPTION:
The symptomatic management of COVID-19 infections is currently at the forefront. The therapeutic efficacy of certain molecules is being evaluated in studies, in vitro and in vivo, such as remdesivir, hydroxychloroquine / chloroquine, and lopinavir / ritonavir. The latter has been used in the treatment of HIV for many years, like other PIs such as darunavir and atazanavir. In France, around 11% of PLWHIV are treated with long-term PIs.

Lopinavir / ritonavir has an inhibitory role on the protein endopeptidase of coronavirus C30 (CEP_C30). In humans, Cao et al did not demonstrate any superiority of efficacy of lopinavir / ritonavir compared to the control group receiving standard care (HR for clinical improvement: 1.24 (0.90-1, 72)), but the initiation of treatment in the study was mainly at late stages. Early initiation of lopinavir/r at the onset of SARS symptoms appears to be more effective. To our knowledge, the other PIs are under study, with a possible inhibition of the proteases of type-3-chemotrypsin or of the papain type of SARS-Cov2. Three open randomized studies in humans are underway in China, Spain, and Thailand. The question arises as to whether treatment with PIs could have a preventive role for COVID-19 infection, especially since PLWHIV have not been described as more at risk of developing COVID-19 infection.

The aim of our study will therefore be to assess the impact of long-term protease inhibitors in PLWHIV on the incidence of COVID-19.

This is a prospective multicenter cohort study. A random sample of 794 eligible individuals will be recruited from April 2020, consisting of 397 patients in the long-term PIs group and 397 patients in the long-term ARV regimen without PIs. The study will be offered to PLWHIV in Île-de-France, treated with long-term antiretroviral drugs with or without protease inhibitors.

For those who accept: i) they will receive phone calls (teleconsultation) to collect information regarding symptoms at M0, M1 and between M3 and M6 by a medical or paramedical person from their hospital center ; ii) in case of a high probability of infection with Covid-19, an on-site consultation will be offered to them, with a diagnostic test by PCR on a nasopharyngeal swab and eventually a chest scanner if indicated ; iii) a serology on a blood sample will be performed at the end of the epidemics to look for anti-COVID-19 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients over 18 years of age
* Follow-up for an HIV infection 1 or 2
* Treated with antiretroviral drugs
* Resident in France during the epidemics
* No change in antiretroviral drugs during the epidemics
* No-opposition to participate to the research

Exclusion Criteria:

* Patients under guardianship or curators
* Opportunistic classifying pathologies by the Control Disease Center (CDC)
* Patients unable to give a free and informed no-opposition consent to participate to the protocol
* Patients under safeguarding justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to HIV patients treated with long-term antiretroviral drugs (ARDs) with or without protease inhibitors (PIs).
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the incidence of COVID-19 infection in PLWHIV treated with long-term antiretroviral drugs including a protease inhibitor and those without a protease inhibitor | 1 month
  Occurrence of COVID-19 infection during the epidemics (M0, M1) in both study groups

SECONDARY OUTCOMES:
Determination of the seroprevalence of COVID-19 infection in both groups of the study | 6 months
  Percentage of positive serological tests at the end of the epidemics in both study groups
Comparison of the severity of COVID-19 infection symptoms in both groups of the study. | 6 months
  Proportion of severe forms in both study groups
Identification of potential risk factors for COVID-19 infection in HIV patients treated with protease inhibitor or without protease inhibitor | 6 months
  Statistical association between a risk factor and the occurrence of COVID-19 infection in both study groups

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHI Créteil, Créteil
  - CHU Henri Mondor, Créteil
  - Centre hospitalier de Melun (GHSIF), Melun
  - Hopital universitaire de Hotel Dieu, Paris
  - Hopital Universitaire de Necker, Paris
  - CHI Villeneuve St Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No